CLINICAL TRIAL: NCT01252667
Title: A Phase II Study of Optimally Dosed Clofarabine in Combination With Low-Dose TBI to Decrease Relapse Rates After Related or Unrelated Donor Hematopoietic Cell Transplantation in Patients With AML
Brief Title: Clofarabine and Low-Dose Total-Body Irradiation in Treating Patients With Acute Myeloid Leukemia Undergoing Donor Peripheral Blood Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2430.00; NCI-2010-02247 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2430.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA078902 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2010-11-29; First posted 2010-12-03 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Cyclosporine; Cyclosporins; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Intervention Model Description: In part 1, patients are treated at each dose in cohorts of three and observed for any dose limiting toxicities. In Part 2, patients are treated at the maximum tolerated dose established in Part 1.
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Part 1 - Dose 1 (30 mg/m^2 Clofarabine) (Experimental): CONDITIONING REGIMEN: Patients receive 30 mg/m^2 clofarabine IV over 2 hours on days -6 to -2. Patients also undergo TBI on day 0.
  IMMUNOSUPPRESSION: Patients with related donors receive cyclosporine PO every 12 hours on days -3 to 56 with taper to day 180 and mycophenolate mofetil PO every 12 hours on days 0 to 28. Patients with unrelated donors receive cyclosporine PO every 12 hours on days -3 to 100 with taper to day 180 and mycophenolate mofetil PO every 8 hours on days 0 to 40 with taper to day 96.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Clofarabine: Given IV
  Cyclosporine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Pharmacological Study: Optional correlative studies
  Total-Body Irradiation: Undergo TBI
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Clofarabine; Drug: Cyclosporine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Radiation: Total-Body Irradiation
- Part 1 - Dose 2 (40 mg/m^2 Clofarabine) (Experimental): CONDITIONING REGIMEN: Patients receive 40 mg/m^2 clofarabine IV over 2 hours on days -6 to -2. Patients also undergo TBI on day 0.
  IMMUNOSUPPRESSION: Patients with related donors receive cyclosporine PO every 12 hours on days -3 to 56 with taper to day 180 and mycophenolate mofetil PO every 12 hours on days 0 to 28. Patients with unrelated donors receive cyclosporine PO every 12 hours on days -3 to 100 with taper to day 180 and mycophenolate mofetil PO every 8 hours on days 0 to 40 with taper to day 96.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Clofarabine: Given IV
  Cyclosporine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Pharmacological Study: Optional correlative studies
  Total-Body Irradiation: Undergo TBI
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Clofarabine; Drug: Cyclosporine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Radiation: Total-Body Irradiation
- Part 1 - Dose 3 (50 mg/m^2 Clofarabine) (Experimental): CONDITIONING REGIMEN: Patients receive 50 mg/m^2 clofarabine IV over 2 hours on days -6 to -2. Patients also undergo TBI on day 0.
  IMMUNOSUPPRESSION: Patients with related donors receive cyclosporine PO every 12 hours on days -3 to 56 with taper to day 180 and mycophenolate mofetil PO every 12 hours on days 0 to 28. Patients with unrelated donors receive cyclosporine PO every 12 hours on days -3 to 100 with taper to day 180 and mycophenolate mofetil PO every 8 hours on days 0 to 40 with taper to day 96.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Clofarabine: Given IV
  Cyclosporine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Pharmacological Study: Optional correlative studies
  Total-Body Irradiation: Undergo TBI
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Clofarabine; Drug: Cyclosporine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Radiation: Total-Body Irradiation
- Part 2 - Dose 1 (30 mg/m^2 Clofarabine) (Experimental): CONDITIONING REGIMEN: Patients receive 30 mg/m^2 clofarabine IV over 2 hours on days -6 to -2. Patients also undergo TBI on day 0.
  IMMUNOSUPPRESSION: Patients with related donors receive cyclosporine PO every 12 hours on days -3 to 56 with taper to day 180 and mycophenolate mofetil PO every 12 hours on days 0 to 28. Patients with unrelated donors receive cyclosporine PO every 12 hours on days -3 to 100 with taper to day 180 and mycophenolate mofetil PO every 8 hours on days 0 to 40 with taper to day 96.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Clofarabine: Given IV
  Cyclosporine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Pharmacological Study: Optional correlative studies
  Total-Body Irradiation: Undergo TBI
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Clofarabine; Drug: Cyclosporine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Radiation: Total-Body Irradiation
- Part 2 - Dose 2 (40 mg/m^2 Clofarabine) (Experimental): CONDITIONING REGIMEN: Patients receive 40 mg/m^2 clofarabine IV over 2 hours on days -6 to -2. Patients also undergo TBI on day 0.
  IMMUNOSUPPRESSION: Patients with related donors receive cyclosporine PO every 12 hours on days -3 to 56 with taper to day 180 and mycophenolate mofetil PO every 12 hours on days 0 to 28. Patients with unrelated donors receive cyclosporine PO every 12 hours on days -3 to 100 with taper to day 180 and mycophenolate mofetil PO every 8 hours on days 0 to 40 with taper to day 96.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Clofarabine: Given IV
  Cyclosporine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Pharmacological Study: Optional correlative studies
  Total-Body Irradiation: Undergo TBI
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Clofarabine; Drug: Cyclosporine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Radiation: Total-Body Irradiation
- Part 2 - Dose 3 (50 mg/m^2 Clofarabine) (Experimental): CONDITIONING REGIMEN: Patients receive 50 mg/m^2 clofarabine IV over 2 hours on days -6 to -2. Patients also undergo TBI on day 0.
  IMMUNOSUPPRESSION: Patients with related donors receive cyclosporine PO every 12 hours on days -3 to 56 with taper to day 180 and mycophenolate mofetil PO every 12 hours on days 0 to 28. Patients with unrelated donors receive cyclosporine PO every 12 hours on days -3 to 100 with taper to day 180 and mycophenolate mofetil PO every 8 hours on days 0 to 40 with taper to day 96.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Clofarabine: Given IV
  Cyclosporine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic hematopoietic PBSCT
  Pharmacological Study: Optional correlative studies
  Total-Body Irradiation: Undergo TBI
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Clofarabine; Drug: Cyclosporine; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoietic PBSCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; allogeneic stem cell transplantation; HSC; HSCT
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic hematopoietic PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; peripheral stem cell support; Peripheral Stem Cell Transplant; peripheral stem cell transplantation
Other: Pharmacological Study — Optional correlative studies
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies the side effects and how well clofarabine works when given together with low-dose total-body irradiation (TBI) in treating patients with acute myeloid leukemia (AML) undergoing donor peripheral blood stem cell transplant (PBSCT). Giving chemotherapy and TBI before a donor PBSCT helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of clofarabine in combination with 2, 3, or 4 Gy TBI in preparation for hematopoietic cell transplantation (HCT) from human leukocyte antigen (HLA)-identical related and HLA-matched unrelated donors in patients with AML. (Part 1)

II. To determine the efficacy of the maximum tolerated dose of clofarabine combined with 2, 3, or 4 Gy TBI in reducing the 6 month relapse rate in patients with AML compared to our historical experience with fludarabine and 2 Gy TBI. A satisfactory improvement will be considered 6 month relapse rate declines from 35% to 20% among high-risk (objective for low risk group terminated August 2014). (Part 2)

SECONDARY OBJECTIVES:

I. Leukemia-free and overall survivals.

II. Non-relapse mortality (NRM) of < 5% at 100 days.

III. Engraftment rate of >= 95%.

IV. Prognostic significance of cytogenetics and genetic markers not detected by traditional karyotype analysis, with special respect to tyrosine kinase receptor mutations (such as fms-like tyrosine kinase 3 [FLT3]), retrovirus-associated deoxyribonucleic acid (DNA) sequences (RAS)- and nucleophosmin gene mutations along with CCAAT/enhancer binding protein, alpha (C/EBP) mutations.

V. Rigorous monitoring for minimal residual/recurring disease by standard morphologic, flow cytometric, and molecular techniques in order to facilitate early intervention.

VI. To evaluate the pharmacokinetics of clofarabine (pharmacokinetic samples discontinued January 2017).

OUTLINE: This is a dose-escalation study of clofarabine.

CONDITIONING REGIMEN: Patients receive clofarabine intravenously (IV) over 2 hours on days -6 to -2. Patients also undergo TBI on day 0.

IMMUNOSUPPRESSION: Patients with related donors receive cyclosporine orally (PO) every 12 hours on days -3 to 56 with taper to day 180 and mycophenolate mofetil PO every 12 hours on days 0 to 28. Patients with unrelated donors receive cyclosporine PO every 12 hours on days -3 to 100 with taper to day 180 and mycophenolate mofetil PO every 8 hours on days 0 to 40 with taper to day 96.

TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.

After completion of study treatment, patients are followed up at 4 months and then every year thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >= 55 years with AML OR patients age < 55 years with AML, who also through pre-existing medical conditions or prior therapy are considered to be at high risk for serious toxicities associated with a conventional, high-dose preparative regimen
* Patients must be in morphologic leukemia-free state (marrow blasts < 5%) without evidence of extramedullary disease within 21 days of HCT
* Only patients with Relapse Risk Score > 0 ("high risk") will be enrolled during Part 1; patients with all Relapse Risk Scores will be enrolled during Part 2 (low risk group terminated August 2014)
* HLA-identical related or HLA-matched unrelated donor available
* A signed informed consent form or minor assent form
* DONOR: FHCRC matching allowed will be grade 1.0 to 2.1: unrelated donors who are prospectively: matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* DONOR: A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion; donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT; if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results
* DONOR: Patient and donor pairs homozygous at a mismatched allele are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* DONOR: Peripheral blood stem cells (PBSC) only will be permitted as a HSC source on this protocol

Exclusion Criteria:

* AML French-American-British (FAB) M3 in first complete remission (CR1)
* Active AML involvement of the central nervous system (CNS) with disease refractory to intrathecal chemotherapy
* Presence of circulating leukemic blasts in the peripheral blood detected by standard morphology
* Patients who are human immunodeficiency virus (HIV)+ (HIV+ patients registered at Fred Hutchinson Cancer Research Center [FHCRC] should be offered treatment on Protocol 1410)
* Fertile men and women unwilling to use contraceptive techniques during and for 12 months following treatment
* Left ventricular ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%); ejection fraction is required if age > 50 years or there is a history of anthracycline exposure or history of cardiac disease; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Diffusion capacity of the lung for carbon monoxide (DLCO) < 40% (corrected), total lung capacity (TLC) < 40%, forced expiratory volume in one second (FEV1) < 40% and/or receiving supplementary continuous oxygen
* The FHCRC principal investigator (PI) of the study must approve enrollment of all patients with pulmonary nodules
* Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bridging fibrosis, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, or symptomatic biliary disease
* Serum creatinine should be within normal limits as specified by institutional guidelines; for patients with serum creatinine > upper limit of normal, a 24-hour creatinine clearance will be performed and should be equal to or more than the lower limit of normal
* Karnofsky score < 60 or Lansky score < 50
* Patients with poorly controlled hypertension and on multiple antihypertensives
* Females who are pregnant or breastfeeding
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers) or those with non-hematologic malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within five years; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* The addition of cytotoxic agents for "cytoreduction" with the exception of tyrosine kinase inhibitors (such as imatinib mesylate), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or Rituxan will not be allowed within three weeks of the initiation of conditioning
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Patients with active bacterial or fungal infections unresponsive to medical therapy
* DONOR: Marrow donors
* DONOR: Donors who are HIV-positive and/or medical conditions that would result in increased risk to the donor filgrastim (G-CSF) mobilization and PBSC collections
* DONOR: Identical twin
* DONOR: Any contraindication to the administration of subcutaneous G-CSF at a dose of 16 mg/kg/day for 5 consecutive days
* DONOR: Serious medical or psychological illness
* DONOR: Pregnant or lactating females
* DONOR: Prior malignancy within the preceding 5 years, with the exception of non-melanoma skin cancers
* DONOR: Children < 12 years old

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - University of Colorado Hospital, Aurora, Colorado
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Result] Krakow EF, Gyurkocza B, Storer BE, Chauncey TR, McCune JS, Radich JP, Bouvier ME, Estey EH, Storb R, Maloney DG, Sandmaier BM. Phase I/II multisite trial of optimally dosed clofarabine and low-dose TBI for hematopoietic cell transplantation in acute myeloid leukemia. Am J Hematol. 2020 Jan;95(1):48-56. doi: 10.1002/ajh.25665. Epub 2019 Nov 8. PMID 31637757
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Started | 3 | 3 | 3 | 0 | 0 | 35
Completed | 3 | 3 | 3 | 0 | 0 | 34
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Transplant aborted post-conditioning | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: No subjects were treated with Dose 1 or 2 in Part 2 as no DLTs were observed in Part 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 35 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  |  | 0 | 0
  Between 18 and 65 years | 0 | 2 | 1 |  |  | 8 | 11
  >=65 years | 3 | 1 | 2 |  |  | 27 | 33
Age, Continuous [Median (Full Range); unit: years] | 73.4 [67.3 to 73.7] | 64.1 [59.9 to 67.1] | 67.7 [53.6 to 68.6] |  |  | 69.5 [54.8 to 74.5] | 69.1 [53.6 to 74.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 |  |  | 13 | 16
  Male | 2 | 2 | 2 |  |  | 22 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 |  |  | 2 | 2
  Not Hispanic or Latino | 3 | 3 | 3 |  |  | 31 | 40
  Unknown or Not Reported | 0 | 0 | 0 |  |  | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  |  | 0 | 0
  Asian | 0 | 0 | 0 |  |  | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  | 0 | 0
  Black or African American | 0 | 0 | 0 |  |  | 0 | 0
  White | 3 | 3 | 3 |  |  | 32 | 41
  More than one race | 0 | 0 | 0 |  |  | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 |  |  | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 |  |  | 35 | 44

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLT)
Description: The primary objective of part 1 is to determined the highest dose of clofarabine that can be tolerated safely in conjunction with nonmyeloablative transplant. If three patients successfully transplant without DLT, dose escalation occurs. If one of those three patients experiences DLT an additional three patients will be treated using the same dose. If a second DLT is observed in the first 3-6 patients, or if three patients are successfully transplanted without DLT at the highest dose the study will proceed to Part 2 using the maximum tolerated dose.
  A Clofarabine related dose-limiting toxicity is defined as a grade 4 toxicity involving the lungs, heart, liver (not resolving in 48 hours), kidneys (not resolving in 48 hours), gastrointestinal tract, and/or central nervous system.
Time Frame: 14 days post-transplant
Population: Analysis only applies to subjects accrued in Part 1 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2: Number of Participants With Relapsed Disease
Description: Number of high risk patients with relapsed disease after receiving the maximum dose of clofarabine. Relapse is defined as the presence of >5% aberrant blasts by morphology on a marrow aspirate or the presence of circulating blasts in the peripheral blood.
Time Frame: 6 months post-transplant
Population: Analysis only applies to subjects accrued in Part 2 of the study. Two subjects in Low Risk status and not evaluable toward this outcome. One subject aborted transplant during conditioning and subsequently expired. This subject was counted towards accrual but not evaluated with respect to outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 32
Participants | 0 | 0 | 0 | 0 | 0 | 3

3. Secondary Outcome: Number of Participants Surviving Progression-free.
Description: Number of patients surviving without progressive disease post-transplant. Progression is defined as the presence of >5% aberrant blasts by morphology on a marrow aspirate or the presence of circulating blasts in the peripheral blood.
Time Frame: 1 Year post-transplant
Population: No subjects were treated with Dose 1 or 2 in Part 2 as no DLTs were observed in Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 35
Participants | 0 | 2 | 1 | 0 | 0 | 21

4. Secondary Outcome: Number of Participants Surviving Overall
Description: Number of patients surviving overall post-transplant.
Time Frame: 1 Year post-transplant
Population: No subjects were treated with Dose 1 or 2 in Part 2 as no DLTs were observed in Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 35
Participants | 0 | 2 | 1 | 0 | 0 | 22

5. Secondary Outcome: Number of Non-Relapse Mortalities (NRM)
Description: Number of patients who expired without disease progression/relapse.
Time Frame: 100 days post-transplant
Population: No subjects were treated with Dose 1 or 2 in Part 2 as no DLTs were observed in Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 35
Participants | 0 | 1 | 0 | 0 | 0 | 1

6. Secondary Outcome: Number of Participants Who Graft Rejected.
Description: Number of patients who graft rejected post-transplant. Graft rejection is defined as <5% donor peripheral blood T cells (CD3+).
Time Frame: 1 Year post-transplant.
Population: No subjects were treated with Dose 1 or 2 in Part 2 as no DLTs were observed in Part 1. One subject on Part 2 Dose 3 aborted transplant during conditioning and subsequently expired. This subject was counted towards accrual but not evaluated with respect to outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 34
Participants | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Prognostic Significance of Cytogenetic and Genetic Markers
Description: Potential prognostic markers will be assessed by polymerase chain reaction (PCR) to determine their prognostic value.
Time Frame: 1 Year post-transplant
Population: The studies have not been carried out on the specimens to evaluate this outcome measure.
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Minimal Residual/Recurring Disease (MRD) Post-transplant
Description: Number of patients with MRD post-transplant, detected in the bone marrow as cytogenetic abnormalities or <5% monoclonal blasts by flow cytometry.
Time Frame: 1 Year post-transplant
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 35
Participants | 0 | 2 | 0 | 0 | 0 | 6

9. Secondary Outcome: Pharmacokinetics (PK) of Clofarabine
Description: Pharmacokinetic measurement of the volume of plasma from which clofarabine is completely removed per unit time. Clearance normalized to actual body weight. Pharmacokinetic analyses were performed on only a subset of patients and no aggregate calculations were made using the data.
Time Frame: Blood was drawn on day -6 before the first clofarabine dosing, at the end of the infusion, and at 3, 4, 5, 6 and 24 hours after the start of infusion. Only pre-dose samples were drawn on days -5, -4, and -3.
Population: Pharmacokinetic analyses were performed on only a subset of patients.
Measure: Number; unit: L/h/kg
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
Number analyzed (Participants) | 0 | 2 | 3 | 0 | 0 | 0
L/h/kg
  ID 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  ID 1 |  | 0.53 |  |  |  |
  ID 2: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  ID 2 |  | 0.37 |  |  |  |
  ID 4: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  ID 4 |  |  | 0.29 |  |  |
  ID 5: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  ID 5 |  |  | 0.40 |  |  |
  ID 6: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  ID 6 |  |  | 0.50 |  |  |

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200; All-Cause Mortality: Conditioning through 1 Year.
Description: No subjects were treated with Dose 1 or 2 in Part 2 as no DLTs were observed in Part 1.
Arm/Group | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine)
All-Cause Mortality (participants affected / at risk) | 3/3 | 1/3 | 2/3 | 0/0 | 0/0 | 13/35
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/0 | 0/0 | 0/35
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 0/0 | 0/0 | 18/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Dose 1 (30 mg/m^2 Clofarabine) (N=3) | Part 1 - Dose 2 (40 mg/m^2 Clofarabine) (N=3) | Part 1 - Dose 3 (50 mg/m^2 Clofarabine) (N=3) | Part 2 - Dose 1 (30 mg/m^2 Clofarabine) (N=0) | Part 2 - Dose 2 (40 mg/m^2 Clofarabine) (N=0) | Part 2 - Dose 3 (50 mg/m^2 Clofarabine) (N=35)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | NA | NA | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | NA | NA | 2 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | 2 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | NA | NA | 3 (3)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Constrictive pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 4 (4)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 3 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 2 (2)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0) | NA | NA | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT01252667/Prot_SAP_000.pdf